CLINICAL TRIAL: NCT00439790
Title: Validation of a Prognostic Score to Identify Heart Failure Patients Who Might Need an Implantable Cardioverter Defibrillator Using Muscle Sympathetic Nerve Activity and Autonomic Testing
Brief Title: Sympathetic Nerve Activity and an Implantable Cardioverter Defibrillator in Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 0602508
Record Dates: First submitted 2007-02-23; First posted 2007-02-26 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: Heart Failure; Death, Sudden, Cardiac
Keywords: implantable cardioverter defibrillator; Heart failure; Sudden Cardiac Arrest; appropriate shock; Defibrillators, Implantable
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Microneurography — Microneurography

SUMMARY:
The aim of this study is to analyze whether the sympathetic tone, measured indirectly and directly by muscle sympathetic nerve activity recording, is elevated in patients with heart failure receiving an appropriate shock from their implantable cardiac defibrillator (ICD) compared to heart failure patients not receiving a shock from their ICD. All parameters measured in this study will be used to build a risk algorithm able to identify heart failure patients at high risk for sudden cardiac death who could receive an ICD.

DETAILED DESCRIPTION:
We plan to perform an extensive study of the sympathetic nervous system activity in heart failure patients with an ICD. The SNS activity will be measured directly by a recording of the muscle sympathetic nerve activity and indirectly by post processing of 24-hour Holter recording, catecholamine levels assessment, and spontaneous baroreflex sensitivity. A global assessment of the patients status will also be realised. Patients will be followed for one year. During follow up, this cohort will be divided into two groups according to the occurrence or not of an appropriate shock. We assume that an appropriate shock is a surrogate marker for sudden cardiac death. We plan to compare the autonomic nervous system activity in both groups of patients in order to identify a score able to detect heart failure patients at high risk for sudden cardiac death.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure patient with an ICD

Exclusion Criteria:

* Pregnant patient
* Acute coronary syndrome within the last 3 months
* Peripheral neuropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patient
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2007-01; Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Pathak, MD, Principal Investigator — Hospital University Toulouse
Locations (1):
- Cardiologie, University Hospital, Toulouse, France